CLINICAL TRIAL: NCT01210365
Title: Safety and Efficacy of the Combination of Furosemide 40 mg + Amiloride Hydrochloride 10 mg in the Reduction of Edema of Cardiac Origin in Patients With Congestive Heart Failure Functional Class II (NYHA)
Brief Title: Safety and Efficacy of Furosemide 40mg + Amiloride Hydrochloride 10mg to Reduct Edema
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: EF decided suspended the study because the investigational product was changed.
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF083
Record Dates: First submitted 2010-08-09; First posted 2010-09-28 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Congestive Heart Failure
Keywords: CHF functional class II; Patients with CHF; Patients with CHF functional class II (NYHA) of any etiology
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- furosemide (40 mg) +amiloride (10 mg) (Experimental): One group of patients will receive furosemide 40 mg + amiloride chloride 10 mg.The patient will swallow the tablet in whole form on an empty stomach with some liquid.
  Interventions: Drug: Diurisa®
- Lasix ® (Active Comparator): One group of patients will receive Lasix® (furosemide 40 mg). For treatment, the patient will swallow the tablet in whole form on an empty stomach with some liquid.
  Interventions: Drug: Lasix ®

INTERVENTIONS:
Drug: Diurisa® — Furosemide 40 mg + amiloride chloride 10 mg.The patient will swallow onde tablet per day in whole form on an empty stomach with some liquid during 4 weeks.
  Arms: furosemide (40 mg) +amiloride (10 mg)
Drug: Lasix ® — One group of patients will receive furosemide 40mg .The patient will swallow the tablet in whole form on an empty stomach with some liquid.
  Arms: Lasix ®

SUMMARY:
The study consists in two treatment groups, one group will receive Diurisa® (furosemide 40 mg + amiloride chloride 10 mg) and the other one will receive furosemide 40 mg (Lasix®)

DETAILED DESCRIPTION:
General Purpose

1. To comparatively evaluate the tolerability and efficacy of a fixed combination of furosemide (40 mg) and amiloride (10 mg) compared with furosemide alone, in the treatment of patients with HF functional class II (NYHA)

Specific Purposes

1. To evaluate the effect on kalemia of the fixed combination of furosemide and amiloride compared with furosemide alone in the treatment of patients with HF functional class II (NYHA)
2. To evaluate the efficacy of the fixed combination of furosemide and amiloride in reducing edema of the LLLL, as compared with furosemide alone, in the treatment of patients with HF functional class II (NYHA).

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years old
2. Must be able to follow instructions and attend study visits.
3. Diagnosis of CHF functional class II (NYHA) without prior use of diuretics
4. Women of childbearing potential who are using a reliable contraceptive method, as assessed by the principal investigator

Exclusion Criteria:

1. Any clinically significant, serious or severe medical condition (e.g., Thyroid, renal or liver disorder, Chronic Obstructive Pulmonary Disease, etc.)
2. History of acute myocardial infarction (within 6 months) or decompensated coronary artery disease
3. Pulmonary hypertension - PASP > 45 mmHg
4. Fasting blood glucose above 150 mg/dl
5. Psychiatric or neurological disorders
6. A condition that, according to Principal Investigator's opinion, may interfere with the optimal study participation or which may put the patient at special risk.
7. Participation in any other investigational study within 12 months before signing the ICF.
8. Known medical history of allergy, hypersensitivity or intolerance to any of the components of the drugs to be used in this study.
9. Any medical treatment that is unrelated to the study and scheduled to the clinical trial period, except for non-serious well-controlled comorbidities which are already being followed up medically.
10. Another drug scheduled to be initiated after study entry.
11. Obesity - BMI > 30 kg/m2
12. Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect on kalemia of the fixed combination of furosemide and amiloride compared with furosemide alone in the treatment of patients with HF functional class II (NYHA) | 5 months
  General physical examination and measure of potassium level in blood will be used for measuring the improvement of CHF symptoms and decrease in peripheral edema. The exams will be performed before the enrollment in the clinical study and every 7 days. Patients who have potassium levels below normal (normal K+ ≥ 3.5 mEq/l) after visit 2 may receive oral replacement, at the investigator's discretion, pursuant to the study site routine. The final evaluation will be performed 42 days after the inclusion of the last patient.

CONTACTS AND LOCATIONS:
Overall Officials: Juliano N Cardoso, Principal Investigator — Casa de Saúde santa Marcelina; Rafael S Silva, Principal Investigator — SITCOR - Assistência Médica Integrada; Luiz Maurino, Principal Investigator — Hospital dos Servidores do Estado - Rio de Janeiro
Locations (4):
- Brazil (4):
  - Centro de Estudos de Diabetes e Hipertensão, Fortaleza, Ceará
  - Hospital dos Servidores do estado - Rio de Janeiro, Rio de Janeiro
  - Casa de Saúde Santa Marcelina, São Paulo
  - SITCOR Assistência Médica Integrada, São Paulo